CLINICAL TRIAL: NCT00918749
Title: Study Assessing the Efficacy, Safety, and Pharmacokinetics of 75 and 100 mg Once-a-month Delayed-release Risedronate Formulations Compared to 150 mg Once-a-month Immediate-release Risedronate for 3 Months in Postmenopausal Women Age 45-80
Brief Title: Delayed Release (DR) Risedronate Compared to Immediate Release (IR) in Postmenopausal Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2009003
Record Dates: First submitted 2009-06-10; First posted 2009-06-11 (Estimated); Results first posted 2011-03-24 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-06

CONDITIONS: Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 150 mg (Active Comparator): 150 mg risedronate tablet IRBB (immediate release before breakfast) administered orally at least 30 minutes before breakfast.
  Interventions: Drug: 150 mg
- 75 mg (Experimental): 75 mg risedronate tablet DRFB (delayed release following breakfast) administered orally immediately after ingesting breakfast
  Interventions: Drug: 75 mg
- 100 mg (Experimental): 100 mg risedronate tablet DRFB (delayed release following breakfast) administered orally immediately after ingesting breakfast
  Interventions: Drug: 100 mg

INTERVENTIONS:
Drug: 150 mg — 150 mg immediate release (IRBB) risedronate tablet administered orally at least 30 minutes before breakfast.
  Arms: 150 mg
Drug: 75 mg — 75 mg delayed release (DRFB) risedronate tablet administered orally immediately after ingesting breakfast
  Arms: 75 mg
Drug: 100 mg — 100 mg delayed release (DRFB) risedronate tablet administered orally immediately after ingesting breakfast
  Arms: 100 mg

SUMMARY:
Randomized, multicenter, double-blind, double-dummy, active-controlled, parallel-design study in approximately 201 postmenopausal women. A subset of subjects (approximately 102) will also participate in a pharmacokinetic (PK) component of the study. Each subject will be randomized to 1 of 3 treatment regimens for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* female, 45 to 80 years of age, in good general health
* postmenopausal ≥2 years, surgically or naturally
* body mass index less than or equal to 32 kg/m^2 at screening

Exclusion Criteria:

* no use within 3 months prior, nor use for more than 1 month at any time within 6 months of: glucocorticoids, anabolic steroids, estrogens, selective estrogen-receptor modulators (SERMs), or estrogen-related drugs, progestins, calcitonin, vitamin D supplements (>1200 IU per day), calcitriol, calcidiol, or alfacalcidol at any dose, any bisphosphonate. fluoride (≥10 mg/day), strontium (≥50 mg/day), parathyroid hormone, investigational bone active agents.
* allergic or abnormal reactions to bisphosphonates
* history of cancer within 5 years, excluding squamous and basal cell carcinoma with 6 month remission
* positive pregnancy test
* no depot injection >10,000 IU vitamin D in previous 9 months.
* no history of GI disease that requires medication, or history of Crohn's disease, ulcerative colitis, diverticular disease, polyps, or surgery that could have changed GI structure or motility.
* no history of frequent diarrhea or constipation that requires regular laxative use.
* no history of alcohol or durg abuse, hyperparathyroidism, cancer previous 5 years, major surgery within 1 month prior to screening, diabetes, uncontrolled hypertension, cardiovascular, hepatic, renal or GI disease.
* no active hyperthyroidism, osteomalacia, use of anticonvulsant medication, or allergic reaction to bisphosphonates

Ages: 45 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2009-05; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chantell Wilson, PhD, Study Director — Procter and Gamble
Locations (6):
- United States (6):
  - Research Site, Daytona Beach, Florida
  - Research Site, Fort Myers, Florida
  - Research Site, Honolulu, Hawaii
  - Research Site, Evansville, Indiana
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Screening began 27 May 2009
Period: Overall Study
Arm/Group | 150 mg | 75 mg | 100 mg
Started | 70 | 66 | 69
ITT (Intent to Treat) Population | 69 (One subject took no study drug and was not included in ITT Population) | 66 | 69
Completed | 63 | 63 | 62
Not Completed | 7 | 3 | 7
Not completed — Adverse Event | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal by Subject | 5 | 3 | 5
Not completed — No Study Medication Taken | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 150 mg | 75 mg | 100 mg | Total
Number analyzed (Participants) | 70 | 66 | 69 | 205
Age, Continuous [Mean (Standard Deviation); unit: years] — ITT Population
  years | 58.3 (7.2) | 58.2 (7.2) | 57.5 (7.0) | 58.0 (7.1)
Age, Customized [Number; unit: participants] — ITT Population - Total 204
  participants
    < 65 years | 57 | 53 | 55 | 165
    65 years thru <75 years | 10 | 12 | 13 | 35
    >= 75 years | 2 | 1 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 66 | 69 | 205
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants] — ITT Population
  Participants
    Asian (Oriental) | 7 | 6 | 3 | 16
    Black | 0 | 4 | 3 | 7
    Caucasian | 60 | 53 | 61 | 174
    Multi-Racial | 1 | 3 | 1 | 5
    Hawaiian/Pacific Islander | 1 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 70 | 66 | 69 | 205

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline Serum Type-1 Collagen C-telopeptide (CTX) 75 mg & 100 mg DRFB Tablet Compared With 150 mg IRBB Tablet, Month 4, ITT Population
Description: Fasting serum Bone turn-over marker specimen assayed by electochemiluminescence.
Time Frame: Month 4
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Percent Change from Baseline
Arm/Group | 150 mg | 75 mg | 100 mg
Number analyzed (Participants) | 70 | 66 | 69
Percent Change from Baseline | -41.235 (2.995) | -44.832 (3.012) | -53.432 (3.025)
Statistical Analysis 1: Comparison: 150 mg vs 75 mg; A two group t-test with a 0.100 one-sided significance level would have 96% power to detect the difference between a risedronate 150 mg IRBB mean, µ1, of -46.000 and a risedronate 75 mg DRFB mean, µ2, of -29.900 (a difference in means of -16.100), assuming that the common SD was 28.000, with sample sizes of 60 per group, respectively. Estimates were based on Study 2005107 (35 mg DR once a week Phase 2 study). The sample size calculation was not adjusted for multiplicity; Test type: Superiority or Other; p = 0.3946, ANOVA; Fixed effects for treatment and center; LS Mean Difference = -3.598, 90% CI 2-sided [-10.568 to 3.372], Standard Error of Mean 4.215
Statistical Analysis 2: Comparison: 150 mg vs 100 mg; Test type: Superiority or Other; p = 0.0045, ANOVA; Fixed effects for treatment and center; LS Mean Difference = -12.197, 90% CI 2-sided [-19.208 to -5.185], Standard Error of Mean 4.241

2. Secondary Outcome: Percent Change From Baseline CTX 150 mg IRBB Tablet Compared With 75 mg & 100 mg DRFB Tablet, Month 2, ITT Population
Time Frame: 2 months
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Percent Change from Baseline
Arm/Group | 150 mg | 75 mg | 100 mg
Number analyzed (Participants) | 69 | 66 | 69
Percent Change from Baseline | -38.407 (3.504) | -33.641 (3.538) | -38.625 (3.547)
Statistical Analysis 1: Comparison: 150 mg vs 75 mg; Test type: Superiority or Other; p = 0.3372, ANOVA; Fixed effects for treatment and center; LS Mean Difference = 4.765, 90% CI 2-sided [-3.421 to 12.952], Standard Error of Mean 4.952
Statistical Analysis 2: Comparison: 150 mg vs 100 mg; Test type: Superiority or Other; p = 0.9650, ANOVA; Fixed effects for treatment and center; LS Mean Difference = -0.218, 90% CI 2-sided [-8.427 to 7.991], Standard Error of Mean 4.966

3. Secondary Outcome: Percent Change From Baseline CTX 150 mg IRBB Tablet Compared With 75 mg & 100 mg DRFB Tablet, Month 3, ITT Population
Time Frame: 3 months
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Percent Change from Baseline
Arm/Group | 150 mg | 75 mg | 100 mg
Number analyzed (Participants) | 69 | 66 | 69
Percent Change from Baseline | -35.591 (3.045) | -35.203 (3.034) | -46.379 (3.077)
Statistical Analysis 1: Comparison: 150 mg vs 75 mg; Test type: Superiority or Other; p = 0.9276, ANOVA; Fixed effects for treatment and center; LS Mean Difference = 0.388, 90% CI 2-sided [-6.670 to 7.447], Standard Error of Mean 4.269
Statistical Analysis 2: Comparison: 150 mg vs 100 mg; Test type: Superiority or Other; p = 0.0133, ANOVA; Fixed effects for treatment and center; LS Mean Difference = -10.787, 90% CI 2-sided [-17.917 to -3.657], Standard Error of Mean 4.313

4. Secondary Outcome: Percent Change From Baseline Urine NTX (Type-1 Collagen Cross-linked N-telopeptide) Comparing Risedronate 150 mg IRBB Tablet With 75 mg & 100 mg DRFB Tablet, Month 2, ITT Population
Description: Urine NTX Bone turnover marker collected after 8 hour fast, 2nd voided urine between 6-9 am assayed by ELISA.
Time Frame: 2 months
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Percent Change from Baseline
Arm/Group | 150 mg | 75 mg | 100 mg
Number analyzed (Participants) | 69 | 66 | 69
Percent Change from Baseline | -15.365 (6.567) | -0.837 (6.631) | -1.150 (6.689)
Statistical Analysis 1: Comparison: 150 mg vs 75 mg; Test type: Superiority or Other; p = 0.1192, ANOVA; Fixed effects for treatment and center; LS Mean Difference = 14.528, 90% CI 2-sided [-0.813 to 29.868], Standard Error of Mean 9.280
Statistical Analysis 2: Comparison: 150 mg vs 100 mg; Test type: Superiority or Other; p = 0.1298, ANOVA; Fixed effects for treatment and center; LS Mean Difference = 14.215, 90% CI 2-sided [-1.230 to 29.659], Standard Error of Mean 9.343

5. Secondary Outcome: Percent Change From Baseline Urine NTX Comparing Risedronate 150 mg IRBB Tablet With 75 mg & 100 mg DRFB Tablet, Month 3, ITT Population
Description: ITT Population
Time Frame: 3 months
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Percent Change from Baseline
Arm/Group | 150 mg | 75 mg | 100 mg
Number analyzed (Participants) | 69 | 66 | 69
Percent Change from Baseline | -21.673 (4.351) | -20.555 (4.326) | -29.066 (4.356)
Statistical Analysis 1: Comparison: 150 mg vs 75 mg; Test type: Superiority or Other; p = 0.8546, ANOVA; Fixed effects for treatment and center; LS Mean Difference = 1.119, 90% CI 2-sided [-8.956 to 11.193], Standard Error of Mean 6.093
Statistical Analysis 2: Comparison: 150 mg vs 100 mg; Test type: Superiority or Other; p = 0.2291, ANOVA; Fixed effects for treatment and center; LS Mean Difference = -7.393, 90% CI 2-sided [-17.522 to 2.737], Standard Error of Mean 6.126

6. Secondary Outcome: Percent Change From Baseline Urine NTX Comparing Risedronate 150 mg IRBB Tablet With 75 mg & 100 mg DRFB Tablet, Month 4, ITT Population
Description: ITT Population
Time Frame: 4 months
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Percent Change from Baseline
Arm/Group | 150 mg | 75 mg | 100 mg
Number analyzed (Participants) | 69 | 66 | 69
Percent Change from Baseline | -13.447 (6.427) | -7.942 (6.464) | -14.360 (6.492)
Statistical Analysis 1: Comparison: 150 mg vs 75 mg; Test type: Superiority or Other; p = 0.5436, ANOVA; Fixed effects for treatment and center; LS Mean Difference = 5.505, 90% CI 2-sided [-9.452 to 20.462], Standard Error of Mean 9.046
Statistical Analysis 2: Comparison: 150 mg vs 100 mg; Test type: Superiority or Other; p = 0.9201, ANOVA; Fixed effects for treatment and center; LS Mean Difference = -0.914, 90% CI 2-sided [-15.959 to 14.132], Standard Error of Mean 9.100

7. Secondary Outcome: Serum Bone Specific Alkaline Phosphatase (BAP) Comparing Risedronate 150 mg IRBB Tablet With 75 mg & 100 mg DRFB Tablet, Month 2, ITT Population
Description: ITT Population
Time Frame: 2 months
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Percent Change from Baseline
Arm/Group | 150 mg | 75 mg | 100 mg
Number analyzed (Participants) | 69 | 66 | 69
Percent Change from Baseline | -5.457 (2.867) | -2.349 (2.895) | -0.615 (2.902)
Statistical Analysis 1: Comparison: 150 mg vs 75 mg; Test type: Superiority or Other; p = 0.4440, ANOVA; Fixed effects for treatment and center; LS Mean Difference = 3.108, 90% CI 2-sided [-3.590 to 9.807], Standard Error of Mean 4.052
Statistical Analysis 2: Comparison: 150 mg vs 100 mg; Test type: Superiority or Other; p = 0.2349, ANOVA; Fixed effects for treatment and center; LS Mean Difference = 4.842, 90% CI 2-sided [-1.874 to 11.559], Standard Error of Mean 4.063

8. Secondary Outcome: Serum BAP Comparing Risedronate 150 mg IRBB Tablet With 75 mg & 100 mg DRFB Tablet, Month 3, ITT Population
Description: ITT Population
Time Frame: 3 months
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Percent Change from Baseline
Arm/Group | 150 mg | 75 mg | 100 mg
Number analyzed (Participants) | 69 | 66 | 69
Percent Change from Baseline | -17.797 (3.087) | -12.831 (3.075) | -12.872 (3.119)
Statistical Analysis 1: Comparison: 150 mg vs 75 mg; Test type: Superiority or Other; p = 0.2527, ANOVA; Fixed effects for treatment and center; LS Mean Difference = 4.966, 90% CI 2-sided [-2.189 to 12.120], Standard Error of Mean 4.327
Statistical Analysis 2: Comparison: 100 mg; Test type: Superiority or Other; p = 0.2613, ANOVA; Fixed effects for treatment and center; LS Mean Difference = 4.926, 90% CI 2-sided [-2.301 to 12.153], Standard Error of Mean 4.371

9. Secondary Outcome: Serum BAP Comparing Risedronate 150 mg IRBB Tablet With 75 mg & 100 mg DRFB Tablet, Month 4, ITT Population
Description: ITT Population
Time Frame: 4 months
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Percent Change from Baseline
Arm/Group | 150 mg | 75 mg | 100 mg
Number analyzed (Participants) | 69 | 66 | 69
Percent Change from Baseline | -20.885 (2.956) | -19.616 (2.973) | -23.710 (2.986)
Statistical Analysis 1: Comparison: 150 mg vs 75 mg; Test type: Superiority or Other; p = 0.7606, ANOVA; Fixed effects for treatment and center; LS Mean Difference = 1.269, 90% CI 2-sided [-5.609 to 8.148], Standard Error of Mean 4.160
Statistical Analysis 2: Comparison: 100 mg; Test type: Superiority or Other; p = 0.5006, ANOVA; Fixed effects for treatment and center; LS Mean Difference = -2.825, 90% CI 2-sided [-9.744 to 4.095], Standard Error of Mean 4.185

ADVERSE EVENTS:
Time Frame: 27 May 2009 thru 23 October 2009, 5 months
Arm/Group | 150 mg | 75 mg | 100 mg
Serious Adverse Events (participants affected / at risk) | 0/69 | 0/66 | 0/69
Other Adverse Events (participants affected / at risk) | 50/69 | 43/66 | 49/69
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 150 mg (N=69) | 75 mg (N=66) | 100 mg (N=69)
Diarrhoea (Gastrointestinal disorders) | 11 (14) | 15 (20) | 15 (18)
Abdominal Pain (Gastrointestinal disorders) | 5 (5) | 16 (18) | 14 (19)
Nausea (Gastrointestinal disorders) | 6 (8) | 6 (9) | 9 (12)
Vomiting (Gastrointestinal disorders) | 3 (3) | 6 (6) | 6 (6)
Constipation (Gastrointestinal disorders) | 4 (5) | 9 (9) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 4 (4) | 5 (6)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 2 (2) | 4 (4)
Flatulence (Gastrointestinal disorders) | 5 (5) | 2 (2) | 3 (3)
Abdominal Distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (3)
Eructation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Abdominal Pain Lower (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 4 (4) | 0 (0)
Abnormal Faeces (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Frequent Bowel Movements (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 7 (9) | 10 (13)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (8) | 2 (3) | 7 (11)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3 (5) | 2 (2) | 5 (8)
Back Pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 6 (6) | 4 (4)
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0) | 3 (3)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 2 (4)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 3 (3) | 2 (3)
Headache (Nervous system disorders) | 20 (24) | 15 (27) | 18 (25)
Dizziness (Nervous system disorders) | 4 (4) | 4 (4) | 2 (2)
Chills (General disorders) | 1 (1) | 5 (6) | 5 (5)
Pain (General disorders) | 6 (7) | 7 (10) | 5 (6)
Pyrexia (General disorders) | 2 (2) | 2 (2) | 5 (5)
Fatigue (General disorders) | 0 (0) | 2 (3) | 3 (3)
Chest Discomfort (General disorders) | 2 (2) | 1 (2) | 0 (0)
Oedema Peripheral (General disorders) | 2 (2) | 0 (0) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (4) | 1 (1)
Oopharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 0 (0) | 3 (3)
Viral Infection (Infections and infestations) | 2 (2) | 3 (3) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 2 (2)
Decreased Appetite (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 2 (2)
Muscle Strain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less